CLINICAL TRIAL: NCT02223871
Title: A Proof-of-concept Study to Assess the Effect of ACT-451840 Against Early Plasmodium Falciparum Blood Stage Infection in Healthy Subjects
Brief Title: Effect of ACT-451840 Against Early Plasmodium Falciparum Blood Stage Infection in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AC-071-102
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Results first posted 2016-08-10 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Healthy Subjects
Keywords: Malaria; ACT-451840
MeSH Terms: conditions — Malaria | interventions — ACT-451840; Artemether; Lumefantrine; Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACT-451840 500 mg (Experimental): All the participants were infected with Plasmodium falciparum parasites (malaria) using malaria-infected human erythrocytes. When the parasitemia reached 1000 counts/mL, all the participants received 500 mg of ACT-451840 as a single oral dose. Compulsory commencement of treatment with Riamet® (artemether-lumefantrine) to ensure complete clearance of any gametocytes, occurred 16 days after ACT-451840 administration (or earlier if required) for all participants. Primaquine was to be administered as a single dose only in participants for whom gametocytes were still identified after administration of Riamet® rescue medication
  Interventions: Drug: ACT-451840:; Other: Plasmodium falciparum-infected human erythrocytes:; Drug: Artemether 20 mg and lumefantrine 120mg combination tablet:; Drug: Primaquine:

INTERVENTIONS:
Drug: ACT-451840: — ACT-451840 500 mg was provided in 100 mL amber glass bottles formulated as a powder for oral suspension. The ACT-451840 suspension was prepared extemporaneously by addition of 25 mL of water and administered orally under fed condition.
Other: Plasmodium falciparum-infected human erythrocytes: — Each participant was inoculated on Day 0 with approximately 1,800 viable Plasmodium falciparum-infected human erythrocytes administered intravenously.
Drug: Artemether 20 mg and lumefantrine 120mg combination tablet: — Rescue treatment to ensure clearance of Plasmodium falciparum comprising six doses of four tablets (total course of 24 tablets) given over a period of 60 hours. Each dose of tablets administered orally was immediately followed by food or drinks rich in fat (e.g., milk).
  Other Names: Riamet®
Drug: Primaquine: — Rescue treatment to ensure clearance of Plasmodium falciparum, to be taken as a single oral 45 mg dose with food only if gametocytes were identified after administration of Riamet® rescue medication.
  Other Names: Primacin™

SUMMARY:
This was a single-center study using induced blood stage malaria infection to characterize the activity of ACT-451840 against early Plasmodium falciparum blood stage infection

DETAILED DESCRIPTION:
The primary objective of the study was to characterize the activity of ACT-451840 administered orally on clearance of Plasmodium falciparum blood stage parasites from the blood in healthy subjects .The inoculum used for blood stage Plasmodium falciparum challenge (BSPC) contained an estimated 1,800 viable parasite-infected erythrocytes diluted into 2 mL of normal saline for injection. Blood was collected for malaria parasitemia assessment by polymerase chain reaction (PCR). Parasitemia ≥ 1,000 parasites/mL indicated that the subjects should be treated with ACT-451840 . If PCR counts were > 5,000 parasites/mL and symptomatic they were dosed within 24 hours. Subsequent PCR blood sampling were performed prior to ACT-451840 dosing and at 2, 4, 8, 12, 16, 20, 24, 30, 36, 48, 60, 72, 84, 96, 120, 144 hours post-dosing and then approximately times per week until 2 consecutive negative samples, until Riamet® rescue treatment and at the final visit.

ELIGIBILITY:
Inclusion Criteria:

* Body weight, minimum 50 kg, body mass index 18-32 kg/m^2.
* Certified healthy by detailed medical history and physical examination.
* Normal vital signs.
* Normal standard 12-lead electrocardiograph (ECG).
* Laboratory parameters within normal range, unless the investigator considered an abnormality to be clinically irrelevant.
* Use a double barrier method of contraception (male condom plus diaphragm or plus intrauterine device or plus hormonal contraceptive by female partner) for at least 14 days prior to the first dose of study drug until 90 days after the last dose.
* Written informed consent prior to undertaking any study procedure.

Exclusion Criteria:

* Any history of malaria.
* Traveled to or lived (>2 weeks) in a malaria-endemic country in the past 12 months or planned travel to a malaria-endemic country during the course of the study.
* Evidence of increased cardiovascular disease risk.
* History of splenectomy.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician or history of a severe allergic reaction, anaphylaxis or convulsions following any vaccination or infusion.
* Presence of current or suspected serious chronic disease.
* Receiving psychiatric drugs or hospitalized within the past 5 years prior to enrollment for psychiatric illness, history of suicide attempt or confinement for danger to self or others.
* Frequent headaches and/or migraine, recurrent nausea, and/or vomiting.
* Known inherited genetic anomaly.
* Presence of acute infectious disease or fever within the 5 days prior to study product administration.
* Evidence of acute illness within 4 weeks prior to screening.
* Significant intercurrent disease.
* Clinically significant disease or condition that might affect drug absorption, distribution or excretion.
* Any investigational product study within the 12 weeks preceding the study.
* Participation in a research study involving blood sampling greater than 450 mL/ unit of blood, or blood donation to a blood bank during the 8 weeks preceding the reference drug dose in the study.
* Subject unwilling to defer blood donations for 6 months.
* Blood donation within 1 month before inclusion.
* Medical requirement for intravenous immunoglobulin or blood transfusions.
* Previous blood transfusion.
* Symptomatic postural hypotension.
* History or presence of alcohol consumption of more than 40 g per day or drug habituation, or any prior intravenous usage of an illicit substance.
* Smoking more than 5 cigarettes or equivalent per day, unable to stop smoking during the study.
* Ingestion of poppy seeds within 24 hours of the screening blood test.
* Excessive consumption of beverages containing xanthine bases.
* Any medication within 14 days before inclusion or within 5 times the elimination half-life of the medication, vaccination within the last 28 days.
* Corticosteroids, anti-inflammatory drugs, immunomodulators or anticoagulants.
* Recent or current therapy with an antibiotic or drug with potential antimalarial activity.
* Subject who, in the judgment of the investigator, was likely to be non-compliant, or unable to cooperate because of a language problem or poor mental development; was in the exclusion period of a previous study; lived alone; who could not be contacted in case of emergency; who was directly involved in conducting the study; who had no good peripheral venous access.
* Positive result on any of the following tests: hepatitis B surface antigen, anti-hepatitis B core antibodies, anti-hepatitis C virus antibodies, anti-human immunodeficiency virus 1 and 2 antibodies.
* Amphetamine, methamphetamines, barbiturates, benzodiazepines, cocaine, methadone, opiates, phencyclidine, tetrahydrocannabinols, tricyclic antidepressants detected in the urine drug screen unless there was an explanation acceptable to the medical investigator.
* Positive alcohol test.
* Pre-existing prolongation of the interval from beginning of the Q wave until end of the T wave corrected according to Bazett's formula (QTcB interval ) and considered clinically significant.
* Family history of sudden death, congenital prolongation of QTc interval, known congenital prolongation of QTc interval, or any clinical condition known to prolong the QTc interval. History of symptomatic cardiac arrhythmias or clinically relevant bradycardia. Electrolyte disturbances.
* ECG abnormalities at screening which in the opinion of the investigator is clinically relevant or will interfere with the ECG analysis.
* History of clinically significant ECG abnormalities.
* Known hypersensitivity to ACT-451840 or any of its excipients or artemether or other artemisinin derivatives, lumefantrine or other aryl aminoalcohols.
* Unwillingness to abstain from consumption of citrus fruits or their juices, as well as all fruit juices from admission to the end of the confinement period.
* Any history or presence of lactose intolerance.
* Ingestion of any drug since the recruitment interview (other than the doses administered in this study) which, in the opinion of the investigator, could compromise the study.
* Ingestion of any drug in the week prior to dosing or during the blood sampling period which, in the opinion of the investigator, could compromise the study.
* Failure to conform to the requirements of the protocol.
* Detection of any drug listed in the protocol in the urine drug screen unless there was an explanation acceptable to the investigator.
* Vital signs outside the reference range and clinically significant.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Lee, Study Director — Actelion
Locations (1):
- Q-Pharm Clinics, Herston, Queensland, Australia

REFERENCES:
- [Background] Marquart L, Baker M, O'Rourke P, McCarthy JS. Evaluating the pharmacodynamic effect of antimalarial drugs in clinical trials by quantitative PCR. Antimicrob Agents Chemother. 2015 Jul;59(7):4249-59. doi: 10.1128/AAC.04942-14. Epub 2015 May 11. PMID 25963983
- [Result] Krause A, Dingemanse J, Mathis A, Marquart L, Mohrle JJ, McCarthy JS. Pharmacokinetic/pharmacodynamic modelling of the antimalarial effect of Actelion-451840 in an induced blood stage malaria study in healthy subjects. Br J Clin Pharmacol. 2016 Aug;82(2):412-21. doi: 10.1111/bcp.12962. Epub 2016 May 11. PMID 27062080

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This proof-of-concept study was conducted in 8 subjects at a single center in Australia. All the subjects were screened from June 6, 2014 to June 23, 2014 and all were enrolled in the study on June 25, 2014 (Study Day 0).
Groups:
- ACT-451840 500 mg: The subjects were infected with Plasmodium falciparum parasites (malaria) using malaria-infected human erythrocytes. When the parasitemia reached 1000 counts/mL, the subjects received 500 mg of ACT-451840 as an oral single dose. Compulsory commencement of treatment with Riamet® (artemether-lumefantrine) to ensure complete clearance of any gametocytes, occurred 16 days after ACT-451840 administration (or earlier if required).
Period: Overall Study
Arm/Group | ACT-451840 500 mg
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- ACT-451840 500 mg: The subjects were infected with Plasmodium falciparum parasites (malaria) using malaria-infected human erythrocytes. When the parasitemia reached 1000 counts/mL, the subjects received 500 mg of ACT-451840 as an oral single dose. Compulsory commencement of treatment with Riamet® (artemether-lumefantrine) to ensure complete clearance of any gametocytes occurred 16 days after ACT-451840 administration (or earlier if required).
Arm/Group | ACT-451840 500 mg
Number analyzed (Participants) | 8
Age, Continuous [Mean (Full Range); unit: Years] | 24.1 [19 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 4
  Indian | 2
  Asian | 1
  Native Hawaiian | 1

OUTCOME MEASURES:

1. Primary Outcome: Drug-specific Parasite Reduction Ratio (PRR48) of ACT-451840 Over 48 Hours Using a Standardized Approach
Description: After the blood stage Plasmodium falciparum challenge (BSPC), malaria parasitemia was measured by polymerase chain reaction (PCR) in regularly collected blood samples.
  The subject-specific and drug-specific parasite reduction rates over a 48 h period (PRR48) were calculated using an objective standardized approach (observed data over 48 h)
Time Frame: 48 hours after study drug administration
Population: Only subjects with appropriate overall fit (p-value of the overall model F-test <0.001) were taken into account (n = 5)
Measure: Mean (95% Confidence Interval); unit: Ratio
Arm/Group | ACT-451840 500 mg
Number analyzed (Participants) | 5
Ratio | 234.5 [130.4 to 422.0]

2. Secondary Outcome: Maximum Plasma Concentration (Cmax) of ACT-451840
Description: Cmax was directly derived from the plasma concentrations-time curves of ACT-451840. Blood samples for pharmacokinetic characterization were drawn at pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 20, 24, 48, 72, 96, and 144 hours post-dose.
Time Frame: From pre-dose to 144 hours after study drug adminsitration
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | ACT-451840 500 mg
Number analyzed (Participants) | 8
ng/mL | 121.7 [90.6 to 163.5]

3. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of ACT-451840
Description: tmax was directly derived from the plasma concentration-time curves of ACT-451840. Blood samples for pharmacokinetic characterization were drawn at pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 20, 24, 48, 72, 96, and 144 hours post-dose.
Time Frame: From pre-dose to144 hours after study drug administration
Measure: Median (Full Range); unit: Hours
Arm/Group | ACT-451840 500 mg
Number analyzed (Participants) | 8
Hours | 4.0 [3.0 to 6.0]

4. Secondary Outcome: Areas Under the Plasma Concentration-time Curve of ACT-451840
Description: Two AUCs were calculated using non-compartmental analysis: AUC(0-t) from pre-dose to last time-point of measure and AUC(0-inf) from pre-dose and extrapolated to infinity.
  Blood samples for pharmacokinetic characterization were drawn at pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 20, 24, 48, 72, 96, and 144 hours post-dose
Time Frame: From pre-dose to144 hours after study drug administration
Measure: Geometric Mean (95% Confidence Interval); unit: ng*h/mL
Arm/Group | ACT-451840 500 mg
Number analyzed (Participants) | 8
ng*h/mL
  AUC(0-t) | 1254.8 [906.8 to 1736.4]
  AUC(0-inf) | 1284.4 [919.6 to 1794.1]

5. Secondary Outcome: Terminal Half-life [t(1/2)]
Description: Blood samples for pharmacokinetic characterization were drawn at pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 20, 24, 48, 72, 96, and 144 hours post-dose
Time Frame: From pre-dose to144 hours after study drug adminsitration
Population: Per protocol set
Measure: Geometric Mean (95% Confidence Interval); unit: Hours
Arm/Group | ACT-451840 500 mg
Number analyzed (Participants) | 8
Hours | 36.4 [30.2 to 43.9]

6. Secondary Outcome: Change From Baseline in Blood Pressure to End of Study (EOS)
Description: Vital signs, including diastolic and systolic blood pressure (DBP/SBP), were measured at each outpatient visit up to 7 days after ACT-451840 administration, every day during confinement or when malaria symptoms were presented and at the end of study visit (EOS). Other measures were performed if required.
Time Frame: Day 28 (EOS)
Measure: Median (Full Range); unit: mmHg
Arm/Group | ACT-451840 500 mg
Number analyzed (Participants) | 8
mmHg
  SBP at baseline (Day 0) | 121.0 [110.0 to 136.0]
  SBP at EOS (Day 28) | 125.5 [117.0 to 139.0]
  Change from Day 0 to Day 28 in SBP | 2.5 [-5.0 to 20.0]
  DBP at baseline (Day 0) | 66.0 [51.0 to 73.0]
  DBP at EOS (Day 28) | 70.5 [57.0 to 75.0]
  Change from Day 0 to Day 28 in DBP | 0.5 [-3.0 to 12.0]

7. Secondary Outcome: Change From Baseline in Body Temperature up to End of Study (EOS)
Description: Body temperature was measured orally
Time Frame: Day 28 (EOS)
Measure: Median (Full Range); unit: Degree Celsius
Arm/Group | ACT-451840 500 mg
Number analyzed (Participants) | 8
Degree Celsius
  Temperature at baseline (Day 0) | 36.3 [36.0 to 36.7]
  Temperature at EOS (Day 28) | 35.9 [35.8 to 36.4]
  Change from Day 0 to Day 28 in temperature | -0.2 [-0.7 to 0.2]

8. Secondary Outcome: Change From Baseline in Respiratory Rate to End of Study (EOS)
Time Frame: Day 28 (EOS)
Measure: Median (Full Range); unit: Breaths/min
Arm/Group | ACT-451840 500 mg
Number analyzed (Participants) | 8
Breaths/min
  Respiratory rate at baseline (Day 0) | 14 [12 to 18]
  Respiratory rate at EOS (Day 28) | 16 [14 to 18]
  Change from Day 0 to Day 28 in respiratory rate | 1.5 [-4 to 4]

9. Post Hoc Outcome: Drug-specific Parasite Reduction Ratio (PRR48) of ACT-451840 Over 48 Hours Using a New Approach
Description: After the blood stage Plasmodium falciparum challenge (BSPC), malaria parasitemia was measured by polymerase chain reaction (PCR) in regularly collected blood samples.
  The subject-specific and drug-specific parasite reduction rates over a 48 h period (PRR48) were calculated following the data-driven method by Marquart et al. (2015), removing potential lag and tail phases prior to log-linear regression modeling.
Time Frame: 48 hours after study drug administration
Population: Only subjects with appropriate overall fit (p-value of the overall model F-test <0.001) were taken into account (n = 8 with the method described by Marquart et al., 2015)
Measure: Mean (95% Confidence Interval); unit: Ratio
Arm/Group | ACT-451840 500 mg
Number analyzed (Participants) | 8
Ratio | 73.6 [56.1 to 96.5]

ADVERSE EVENTS:
Time Frame: From baseline to end of study
Description: None of the treatment-emergent advserse events reported below were considered related to ACT-451840, one (nausea) was related to Riamet, and all the other ones were related to malaria inoculum
Groups:
- ACT-451840 500 mg: The eight subjects were infected with Plasmodium falciparum parasites (malaria) using malaria-infected human erythrocytes on Day 0 and received 500 mg of ACT-451840 on Day 7. All of them received six doses of Riamet® (artemether-lumefantrine) to ensure complete clearance of any gametocytes, as per protocol.
Arm/Group | ACT-451840 500 mg
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACT-451840 500 mg (N=8)
Pyrexia (General disorders) | 5 (5)
Injection site erythema (General disorders) | 1 (2)
Malaise (General disorders) | 1 (1)
Pain injection site (General disorders) | 3 (3)
Rigors (General disorders) | 1 (1)
Vessel puncture site pain (General disorders) | 1 (1)
Headache (Nervous system disorders) | 7 (10)
Lethargy (Nervous system disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Lip ulcer (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Upper respiratory tract infection (not otherwise specified) (Infections and infestations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Rhesus antibodies positive (Investigations) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the data is under the responsibility of Actelion Pharmaceuticals Ltd. The PI has the opportunity to review the analysis of the data and to discuss with the sponsor the interpretation of the study results prior to publication.